CLINICAL TRIAL: NCT04249297
Title: Multicenter Open-Label Observational Program to Research on Predictors of Pregnancy Rate in Assisted Reproductive Technology in the Russian Population and Kazakhstan Population According to Actual International and National Guidelines (IRIS)
Brief Title: Predictors of Pregnancy Rate in Assisted Reproductive Technology According to Actual Guidelines
Acronym: IRIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: DYDR5005
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Infertility
Keywords: dydrogesterone; Duphaston; Assisted Reproductive Technology; In-Vitro Fertilization; luteal phase support
MeSH Terms: conditions — Infertility | interventions — Dydrogesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IVF/Dydrogesteron: Females aged ≥ 18 years, underwent In-Vitro Fertilization with Elective single embryo transfer in fresh cycle, for whom were prescribed treatment with Duphaston® for luteal phase support as part of an Assisted Reproductive Technology
  Interventions: Drug: Duphaston® (Dydrogesteron)

INTERVENTIONS:
Drug: Duphaston® (Dydrogesteron) — No intervention. Description of routine practice only. Prescribed Duphaston® according local marketing authorization and international and Russian In-Vitro Fertilization guidelines for luteal phase support as part of an Assisted Reproductive Technology (1 tablet 3 times a day starting at the day of oocyte retrieval).

SUMMARY:
Goals: To explore the association of probability of pregnancy with certain prognostic factors in patients undergoing assisted reproductive technology in Russian population according to international and national guidelines.

DETAILED DESCRIPTION:
Research on significant factors (predictors) of pregnancy rate in In Vitro Fertilization (IVF) and Intracytoplasmatic Sperm Injection (ICSI) cycles in Russian population according to actual national and international guidelines in patients using oral dydrogesterone for luteal phase support in assisted reproductive technology. Investigating the strength of the relationship and assessing coefficients of impact on the pregnancy rate.

Creating a predictive table of Clinical Pregnancy in IVF and ICSI cycles and 4-5 most impact predictors.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years
* Prescribed Duphaston® according local marketing authorization and international and Russian In Vitro Fertilisation guidelines for luteal phase support as part of an Assisted Reproductive Technologies (1 tablet 3 times a day starting at the day of oocyte retrieval)
* Elective single embryo transfer in fresh cycle
* Normal ultrasound at enrollment without evidence of clinically significant abnormality consistent with finding adequate for Assisted Reproductive Technologies with respect to uterus and adnexa (incl. no hydrosalpinx or clinically relevant uterine fibroids)
* Signed the Patient Authorization for Use/Disclosure of Data

Exclusion Criteria:

* Evidence of cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurologic/psychiatric, allergy, recent major surgery (< 3 months), or other relevant diseases as revealed by history, physical examination and/or laboratory assessments which could limit participation in or completion of the study
* Acute urogenital disease
* Known allergic reactions to dydrogesterone or other progestogens products
* Any contraindication or other condition that precludes use of dydrogesterone in a particular patient, in accordance with the precautions listed in the locally approved label (Instructions for the medical use of Duphaston®):
* Hypersensitivity to dydrogesterone or any of the excipients
* Diagnosed or suspected progestogen-dependent neoplasms (e.g., meningioma)
* Undiagnosed vaginal bleeding
* Hepatic impairment associated with acute or chronic, current or past liver diseases (as long as liver function tests have failed to return to normal)
* Presence or history of malignant liver tumors
* Galactose intolerance, lactase deficiency, glucose-galactose malabsorption syndrome
* Breastfeeding.
* Presence or history of porphyria
* Age below 18 years, since safety and efficacy in adolescents aged below 18 years have not been established
* Spontaneous abortion (miscarriage) or missed abortion in luteal-phase support as part of assisted reproductive technology
* Participation in any other clinical trial within 30 days prior to program start
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subjects in or to complete the study
* Current or recent substance abuse, including alcohol and tobacco (Note: Patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed)
* History of prior chemotherapy
* Usage of other progestogens except dydrogesterone
* Contraindication for pregnancy
* Refusal or inability to comply with the conditions of this program for any reason, including scheduled clinic visits and laboratory tests.
* Gestational surrogacy, oocyte or embryo donation

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females aged ≥ 18 years, underwent In-Vitro Fertilization with Elective single embryo transfer in fresh cycle, for whom were prescribed treatment with Duphaston® for luteal phase support as part of an Assisted Reproductive Technology
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
4-5 predictors with highest impact on the probability of clinical pregnancy as evaluated by a logistic regression model | 10 weeks
  Evaluating coefficients of the relationship between pregnancy rate and following variables:
  * female age (years),
  * female height (cm) / weight (kg) / Body Mass Index (kg/m2),
  * Antral Follicle Count,
  * Ovarian Sensitivity Index,
  * number of top-quality embryos,
  * pre-implantation genetic testing (performed / not performed),
  * day of embryo transfer,
  * treatment history (number of previous attempts),
  * infertility cause (male factor infertility, endometriosis, endometrial factor, myoma, tubal factor, idiopathic),
  * endometrial thickness,
  * serum Anti-Mullerian hormone level,
  * year, season,
  * race (Caucasian, Asian, Black) as predictors.

SECONDARY OUTCOMES:
Patient's convenience and global satisfaction | 2 weeks, 10 weeks
  Patient's convenience and global satisfaction of using medication for luteal phase support assessed by Treatment Satisfaction Questionnaire for Medication (TSQM-9). TSQM-9 is a 9-item instrument consisting of 3 scales: effectiveness scale (3 questions), convenience scale (3 questions) and global satisfaction scale (3 questions). The scores were computed by adding items for each domain. The lowest possible score was subtracted from this composite score and divided by the greatest possible score minus the lowest possible score. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
The overall pregnancy rate | 10 weeks
  The overall pregnancy rate with confirmed clinical pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs, including ectopic pregnancy
The rate of positive biochemical pregnancy test | 2 weeks
  The rate of positive biochemical pregnancy test (diagnosed by the detection of human chorionic gonadotropin (hCG) in serum or urine on Day 12-14 after embryo transfer).

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana A Nazarenko, Prof, Study Chair — Kulakov National Medical Research Center of Obstetrics, Gynecology and Perinatology
Locations (52):
- Kazakhstan (2):
  - LLP Institute of Reproductive Medicine, Almaty
  - PERSONA International Clinical Center for Reproductology, Almaty
- Russia (50):
  - Regional Clinical Perinatal Center "Dar", Barnaul
  - Clinic of Family Medicine, Chelyabinsk
  - Regional Perinatal Center, Chelyabinsk
  - ART Department Irkutsk Regional Clinical Hospital, Irkutsk
  - Mother and Child, Irkutsk
  - Ivanovo Research Institute motherhood and childhood named after VN Gorodkov, Ivanovo
  - Mother and Child, Kazan'
  - Scandinavia, Kazan'
  - Clinic for male and female health 'OXY-center', Krasnodar
  - Clinic of Kuban State Medical University, Krasnodar
  - Regional Center for Family Health and Reproduction, Krasnodar
  - Mother and Child, Krasnoyarsk
  - IVF Center, Lipetsk
  - Reproductive Health Clinic 'Biootpima', Moscow
  - Generation NEXT, Moscow
  - Medical Center Altra Vita, Moscow
  - Kulakov National Medical Research Center of Obstetrics, Gynecology and Perinatology, Moscow
  - Family Planning and Reproduction Center, Moscow
  - Mother and Child Perinatal Center, Moscow
  - NOVA Clinic, Center for Reproduction and Genetics, Moscow
  - Medical Center MIRA, Moscow
  - Mother and Child Kuntsevo, Moscow
  - Center of Reproduction 'Line of Life', Moscow
  - Mother and Child Savelovskaya, Moscow
  - Clinic 'IVF Center', Moscow
  - Mother and Child Khodynka, Moscow
  - Multidisciplinary Medical Center 'MAK IVF', Moscow
  - Mother and Child Lapino, Moscow
  - Volga Regional Medical Center, Clinical Hospital #1, Nizhny Novgorod
  - Clinical Hospital 'Avicenna', Novosibirsk
  - Novosibirsk Center for Reproductive Medicine 'Mother and Child', Novosibirsk
  - Reproduction Clinic ' Philosophy of Life', Perm
  - Center for Reproductive Technologies 'EmbryLife', Saint Petersburg
  - Ava-Peter Reproduction Clinic, Saint Petersburg
  - Scandinavia Reproduction Clinic, Saint Petersburg
  - Reproductive Medicine Clinic ICLINIC, Saint Petersburg
  - Center for Reproductive Medicine, Saint Petersburg
  - Ott Research Institute of Obstetrics, Gynecology and Reproductology, Saint Petersburg
  - Mother and Child St. Petersburg, Saint Petersburg
  - Mother and Child, Samara
  - Regional Center for Reproductive Medicine Dynasty, Samara
  - Saratov Regional Perinatal Center, Saratov
  - Stavropol Regional Clinical Diagnostic Center, ART Department, Stavropol
  - Center ART, Siberian State Medical University, Tomsk
  - Mother and Child, Tyumen
  - Volgograd State Medical University, Clinik #1, Volgograd
  - Voronezh Regional Clinical Hospital #1, Perinatal Center, Voronezh
  - Research Institute for the Protection of Maternity and Infancy, Yekaterinburg
  - Clinical diagnostic center "Maternal and child health", Yekaterinburg
  - IVF Center Partus, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No